CLINICAL TRIAL: NCT04786301
Title: Severe Acute Respiratory Infection - Preparedness
Brief Title: Severe Acute Respiratory Infection - Preparedness (COVID-19 and Influenza)
Acronym: SARI-PREP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura Evans, Associate Professor, Pulmonary, Critical Care and Sleep Medicine, University of Washington
Other Study IDs: STUDY00011343
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Pneumonia, Viral
MeSH Terms: conditions — Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Severe Acute Respiratory Infection (SARI) is defined by the World Health Organization (WHO) as acute respiratory infection with a history of fever ≥38°C and cough for less than 10 days duration that requires hospital admission. SARI-PREP is a multi-center consortium funded by the CDC Foundation being assembled with the goal of providing the infrastructure to rapidly collect prospective data on clinical risks and outcomes, hospital-level stress, and biologic specimens that will aid in the rapid development of diagnostic and treatment approaches. A current example of a form of SARI to be targeted by SARI-PREP is COVID-19 the acute respiratory infectious disease caused by SARS-CoV-2 infection. COVID-19 has a broad set of manifestations and severity with a subset of affected patients developing severe disease leading to respiratory failure and other forms of organ dysfunction. As with many outbreaks of novel viral pathogens causing SARI there was no efficacious therapeutic intervention at the beginning of the COVID-19 pandemic. Furthermore, while there is emerging knowledge of clinical risks for severe COVID-19, there remains a paucity of information about the viral dynamics and host responses that might indicate a patient is at high risk for poor outcomes.

The COVID-19 pandemic will be the initial target of the SARI-PREP consortium with the overall goal of developing a multi-institutional collaborative network of Acute Care Hospitals that will rapidly enroll, sample, and follow patients admitted with severe COVID-19 and to develop research protocols to rapidly determine demographic, clinical, host molecular, virologic, and institutional correlates of outcome. Overall, the information gained from this effort will help to rapidly inform and improve clinical management of epidemic/pandemic SARI patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission to an acute care or intensive care unit with a clinical syndrome of lower respiratory tract infection suspicious for viral SARI:
* fever
* cough
* AND (radiographic infiltrates by imaging (chest x-ray, CT scan, etc.) OR SpO2 ≤ 94% on room air OR requiring new supplemental oxygen (above baseline if preexisting) OR requiring invasive or non-invasive mechanical ventilation).
* confirmed viral cause for SARI by respiratory viral RT-PCR testing.

Exclusion Criteria:

* Prisoners or wards of the state
* Inability to consent or lack of availability of legal surrogate
* Do not attempt resuscitation/do not intubate status on admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to the hospital with a diagnosis of severe acute respiratory infection.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days (VFD) | 30 days
  Number of days alive and free of mechanical ventilation

SECONDARY OUTCOMES:
Mortality | 28-day and 90-day
Organ failure free days | 30 days
World Health Organization respiratory failure ordinal score | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Laura Evans, MD, MSc, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - NYU Langone Medical Center, New York, New York